CLINICAL TRIAL: NCT04868214
Title: Multi-site Study for Evaluation of Clinical Ranges of Whole Blood Clotting Times of Patients on Anticoagulants and Verification of Measurement Precision of Liquid Quality Controls With the Perosphere Technologies' PoC Coagulometer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sciema UG (Other)
Collaborators: Perosphere Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-01-02-001
Record Dates: First submitted 2021-03-30; First posted 2021-04-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Coagulation
Keywords: coagulation; Factor Xa
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: coagulation measurements — peak and trough coagulation measurements of patients treated with Xarelto, Eliquis, or Lixiana and coagulation measurements of healthy proband blood spiked with eiter Xarelto, Eliquis or Lixiana.

SUMMARY:
The Perosphere Technologies' PoC Coagulometer measures clotting times of fresh whole blood samples. Clotting is initiated by glass surface activation and terminates on optical detection of fibrin assembly, the final step in the coagulation cascade. Since activation occurs at the top of the intrinsic pathway and detection occurs at the bottom of the final common pathway, the Perosphere Technologies' PoC Coagulometer has shown sensitivity to a broad range of drugs and reagents that affect blood clotting processes, including the Direct Oral Anticoagulants, DOACs (e.g. rivaroxaban, apixaban, and edoxaban), as well as the heparins (e.g. enoxaparin, a low molecular weight heparin, and unfractionated heparin). The purpose of the present study is to characterize the performance of the PoC Coagulometer measuring Clotting Time Controls, as well as fresh whole blood from both healthy volunteers and DOAC patients at three field testing sites.

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.
* Be 18- to 80-years-of-age, inclusive, at time of consent.
* Have suitable venous access for at least a single venipuncture.
* Healthy volunteers must: Not be on medication designed to alter the coagulation state of a patient (including anticoagulants, anticoagulant reversal agents, platelet inhibitors, NSAIDs and thrombolytics or "clot buster" drugs), except as specified for phase 3 of testing.
* Eligible patients on anticoagulants must: Have taken their prescribed anticoagulant regularly at least for a month prior to study participation for inclusion in phase 3 of testing
* Eligible patients on anticoagulants must: Have been on their anticoagulant therapy for at least one month.

Exclusion Criteria:

* Have any of the following findings at Study Enrollment (information will be collected via questionnaire): Positive pregnancy test (females); Drug- or alcohol abuse; Use of tobacco or nicotine-containing products within 3 months prior to screening
* Have a personal or family history of clotting disorder or hematologic abnormality, such as excessive bleeding, joint hematoma, thrombovascular disease, thrombocytopenia, or any chronic condition requiring treatment with transfusions.
* Have a history of unexplained syncope.
* Have a history within 6 months prior to Screening of major bleeding, trauma, surgical procedure of any type, or vaginal delivery.
* Have a history within 6 months prior to Screening of peptic ulcer or gastrointestinal bleeding (including hematemesis, melena, or rectal bleeding).
* Have received any blood product or anticoagulant within 3 months prior to Screening.
* Have donated blood or blood products within 3 months prior to Screening.
* Have a history of minor bleeding episodes (e.g., epistaxis, bruising or gingival bleeding) within 1 month prior to screening, or a long-standing history of such bleeding.
* If female, have a history of excessive or dysfunctional uterine bleeding (unless the subject had a subsequent hysterectomy).
* If female, be pregnant, breastfeeding, or planning to become pregnant during the study.

Eligible patients on anticoagulants must not:

* Have a personal or family history of clotting disorder or hematologic abnormality, such as excessive bleeding, joint hematoma, thrombovascular disease, thrombocytopenia, or any chronic condition requiring treatment with transfusions, other than the condition for which a DOAC was prescribed.
* Have a history of unexplained syncope.
* Have a history within 6 months prior to Screening of peptic ulcer or gastrointestinal bleeding (including hematemesis, melena, or rectal bleeding).
* Consume more than 5 cigarettes per day.
* If female, have a history of excessive or dysfunctional uterine bleeding (unless the subject had a subsequent hysterectomy).
* If female, be pregnant, breastfeeding, or planning to become pregnant during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients on rivaroxaban, apixaban, or edoxaban and healthy volunteers between the ages of 18 and 80 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Clotting times of whole blood samples, measured on Perosphere Technologies' PoC Coagulometer devices | During the first/single study visit
  Clotting times measured on Perosphere Technologies´ PoC of patients on Xarelto, Eliquis or Lixiana

SECONDARY OUTCOMES:
Drug concentrations in collected blood samples as measured through anti-factor Xa (anti-Xa) assay | During the first/single study visit
  Drug concentrations in collected blood samples as measured through anti-factor Xa (anti-Xa) assay

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Perosphere Technologies Inc., Danbury, Connecticut
  - Perosphere Technologies Inc., Boynton Beach, Florida
  - Perosphere Technologies Inc., Rockville, Maryland
  - Perosphere Technologies Inc., White Plains, New York
- Pfuetzner Science and Health Institute GmbH, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared